CLINICAL TRIAL: NCT05099614
Title: Naloxone Administration Via Auto-injection in Healthy Volunteers
Brief Title: Naloxone Auto-injection in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jacob Sunshine, Associate Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00005944; 1914873 (Other Grant/Funding Number: NSF)
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Overdose Antidote

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy adults (Experimental): Healthy adults will receive 1.2 mg of naloxone hydrochloride injection solution, administered once via a wearable auto-injector, West Pharma SmartDose Generation I system. The respiratory sensing system under study is used to detect slowed breathing for the purpose of triggering the administration of the naloxone.
  Interventions: Combination Product: Naloxone hydrochloride injection solution, SmartDose wearable auto injector and mobile respiratory sensing system

INTERVENTIONS:
Combination Product: Naloxone hydrochloride injection solution, SmartDose wearable auto injector and mobile respiratory sensing system — 1.2 mg of naloxone hydrochloride is administered to healthy adults using the SmartDose wearable auto injector and the mobile respiratory sensing system.

SUMMARY:
This study continues the work to develop a mobile breathing monitoring system to detect slowed breathing and overdose events caused by opioid use. This is a single-site feasibility study designed to test the mobile application with a commercially available drug delivery device called the SmartDose by West Pharmaceuticals, Inc. The SmartDose is a wearable self-injection device that can deliver a drug under the skin with a push of a button. Naloxone is a drug used to reverse the effects of opioid drugs in the body. This study will evaluate if the mobile application can wireless trigger the delivery of a small dose of naloxone to a healthy adult volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female volunteers
* >18 years
* No allergy to naloxone or ingredients in its formulation
* Ability to read and understand English
* Written informed consent obtained from subject
* Ability to comply with study requirements

Exclusion Criteria:

* History of alcohol or substance abuse
* History of unusual pain sensitivity, lack of sensitivity
* History of chronic myofascial, inflammatory, neuropathic pain
* Chronic use of medication known to interfere with naloxone
* Pregnant women and nursing mothers
* Presence of a condition or abnormality that in the opinion of the Principal Investigator would compromise subject safety or the quality of the data (e.g., persons with liver disease, renal insufficiency/failure)
* Alcohol on the breath

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Detection of slowed breathing that triggers the successful actuation of the auto-injector | The participant breathes to 8 breaths per minute and the breath hold (15 - 30 seconds) triggers the auto-injector. This will take place over 1 -3 minutes.
  Ability of the accelerometer-based system to detect slowed breathing and trigger the successful auto injection of medication
Plasma concentration of naloxone in blood samples | Blood sampling at 3 and 8 minutes after the auto injector is triggered
  The concentration of naloxone in the plasma is measured by blood at two time points

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sunshine, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No